CLINICAL TRIAL: NCT01440140
Title: An Open-label, Three-centre, Randomised, Two-period, Crossover Study to Assess the Efficacy, Safety and Utility of Real-time Continuous Subcutaneous Glucose Monitoring Combined With Overnight Closed-loop Glucose Control in the Home Setting in Comparison With Real-time Continuous Subcutaneous Glucose Monitoring Alone in Adults With Type 1 Diabetes on Subcutaneous Insulin Infusion Pump Therapy
Brief Title: Closing the Loop in Adults With Type 1 Diabetes in the Home Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Principal Investigator, Hood Thabit, Clinical Investigator, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANGELA03
Record Dates: First submitted 2011-09-20; First posted 2011-09-26 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed loop (algorithm) (Experimental)
  Interventions: Other: Closed-loop
- Open loop (Placebo Comparator)
  Interventions: Other: Conventional insulin pump delivery

INTERVENTIONS:
Other: Closed-loop — Subcutaneous delivery of Novorapid insulin, dose calculated by control algorithm, based on continuous glucose sensor readings.
  Other Names: Automated CL
  Arms: Closed loop (algorithm)
Other: Conventional insulin pump delivery — Subcutaneous delivery of Novorapid insulin according to usual pump regime
  Arms: Open loop

SUMMARY:
The main study objective is to compare real-time continuous subcutaneous glucose monitoring (CGM) combined with overnight automated closed-loop glucose control, and real-time CGM alone in the home setting.

DETAILED DESCRIPTION:
Achievement of tight glycaemic control in type 1 diabetes mellitus (T1D) using intensive insulin regimens, which has been shown to be important for the prevention of long term diabetes-related complications, is limited by a significantly increased risk of hypoglycaemia. The average patient with T1D suffers two symptomatic episodes of hypoglycaemia per week, and one episode of severe hypoglycaemia, defined as an event requiring assistance of another person to administer rescue treatment in the form of carbohydrate and/or glucagon, per year.Despite the rapid advancements in insulin pump technology and the ongoing development of more physiological insulin preparations, the currently available therapeutic regimens are still unable to achieve optimal glycaemic control.The emergence of continuous glucose monitoring (CGM) over the last decade, which enables users to view in real-time estimates of plasma glucose and receive alarms for impending hypo- or hyperglycaemia, thus facilitating appropriate changes in insulin therapy, is a major step towards improved diabetes monitoring.

The desirable goal is the development of an insulin delivery that is glucose responsive and the development of effective real time glucose monitoring should allow this. Glucose responsive insulin delivery should allow achievement of ideal glucose targets with less risk of hypoglycaemia. Closed-loop systems may provide a realistic treatment option for people with T1D. The research we are conducting at the University of Cambridge has been focused on developing a closed-loop system for overnight glucose control in patients with T1D. The studies that have been performed so far employ model predictive control (MPC) - this algorithm estimates patient-specific parameters from CGM measurements taken every 1 to 15 minutes and makes predictions of glucose excursions, which are then used to calculate basal insulin infusion rates. We hypothesize that overnight automated closed-loop glucose control in the home setting will be efficacious and safe compared to CGM alone, in T1D subjects on insulin pump treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes, as defined by WHO for at least 6 months or confirmed C-peptide negative.
* On insulin pump therapy for at least 3 months

Exclusion Criteria:

* Non-type 1 diabetes mellitus
* Any physical/psychological disease likely to interfere with the study
* Taking medication likely to interfere with interpretation of the results
* Known/suspected allergy against insulin
* Patients with clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator
* Ongoing severe recurrent hypoglycaemia as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of CGM (Continuous glucose monitoring) values in target (3.9 - 8.0 mmol/l). | 4 weeks
  Participants will be assessed overnight (00:00 to 07:00) for 4 weeks in each arm.

SECONDARY OUTCOMES:
Percentage of CGM values below 3.9 mmol/l. | 4 weeks
  Participants will be assessed overnight (00:00 to 07:00) for 4 weeks in each arm.
Time spent with glucose levels below 3.9 mmol/l and above 8.0 mmol/l, as recorded by CGM and other CGM-based metrics | 4 weeks
  Participants will be assessed overnight (00:00 to 07:00) for 4 weeks in each arm.
Glycaemic control assessed by fructosamine and HbA1c | 4 weeks
  Participants will be assessed for 4 weeks in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, MSc, BSc, Principal Investigator — University of Cambridge
Locations (3):
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - King's College London, London
  - Northern General Hospital, Sheffield

REFERENCES:
- [Derived] Thabit H, Elleri D, Leelarathna L, Allen J, Lubina-Solomon A, Stadler M, Walkinshaw E, Iqbal A, Choudhary P, Wilinska M, Barnard K, Heller S, Amiel S, Evans M, Dunger D, Hovorka R. Unsupervised overnight closed loop insulin delivery during free living: analysis of randomised cross-over home studies in adults and adolescents with type 1 diabetes. Lancet. 2015 Feb 26;385 Suppl 1:S96. doi: 10.1016/S0140-6736(15)60411-1. PMID 26312919
- [Derived] Thabit H, Leelarathna L, Wilinska ME, Elleri D, Allen JM, Lubina-Solomon A, Walkinshaw E, Stadler M, Choudhary P, Mader JK, Dellweg S, Benesch C, Pieber TR, Arnolds S, Heller SR, Amiel SA, Dunger D, Evans ML, Hovorka R. Accuracy of Continuous Glucose Monitoring During Three Closed-Loop Home Studies Under Free-Living Conditions. Diabetes Technol Ther. 2015 Nov;17(11):801-7. doi: 10.1089/dia.2015.0062. Epub 2015 Aug 4. PMID 26241693
- [Derived] Thabit H, Lubina-Solomon A, Stadler M, Leelarathna L, Walkinshaw E, Pernet A, Allen JM, Iqbal A, Choudhary P, Kumareswaran K, Nodale M, Nisbet C, Wilinska ME, Barnard KD, Dunger DB, Heller SR, Amiel SA, Evans ML, Hovorka R. Home use of closed-loop insulin delivery for overnight glucose control in adults with type 1 diabetes: a 4-week, multicentre, randomised crossover study. Lancet Diabetes Endocrinol. 2014 Sep;2(9):701-9. doi: 10.1016/S2213-8587(14)70114-7. Epub 2014 Jun 16. PMID 24943065